CLINICAL TRIAL: NCT03653351
Title: Enhancing Cognition in Older Persons: A Randomized Controlled Trial of Mindfulness-Based Stress Reduction (MBSR) and Transcranial Direct Current Stimulation (tDCS).
Brief Title: Brain Stimulation and Enhancing Cognition in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Eric Lenze, Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID#201805097
Record Dates: First submitted 2018-07-25; First posted 2018-08-31 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Cognitive Impairment, Mild; Depressive Symptoms; Anxiety
MeSH Terms: conditions — Cognitive Dysfunction; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham tDCS and MBSR (Sham Comparator): Includes a combination of 8 weeks of in-class group MBSR + sham tDCS and daily at home MBSR + sham tDCS.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)
- Active tDCS and MBSR (Active Comparator): Includes a combination of 8 weeks of in-class group MBSR + active tDCS and daily at home MBSR + active tDCS.
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation (tDCS) — Transcranial Direct Current Stimulation (tDCS) is a form of neurostimulation (also known as neuromodulation) where very low levels of direct electrical current are delivered to specifically targeted areas of the brain, in order to increase neuroplasticity. The direct current in active tDCS will be of 2 mA (current density = 0.57 A/m2) and will be applied for approximately 30 minutes per day during meditative practices of the MBSR protocol.
  Arms: Active tDCS and MBSR
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Transcranial Direct Current Stimulation (tDCS) is a form of neurostimulation (also known as neuromodulation) where very low levels of direct electrical current are delivered to specifically targeted areas of the brain, in order to increase neuroplasticity. The direct current in active tDCS will be of 2 milliampere (mA) (current density = 0.57 A/m2), however, the device is pre-programmed to turn off after 1 minute of active stimulation (and then turn back on briefly at the end of the 30 minutes).
  Arms: Sham tDCS and MBSR

SUMMARY:
The aim of the current research is to evaluate the efficacy of a combination of Mindfulness-Based Stress Reduction (MBSR) and transcranial direct current stimulation (tDCS) to improve cognitive function in individuals with anxiety, depression and/or cognitive complaints.

DETAILED DESCRIPTION:
Neurocognitive difficulties are a common problem in the older adult population. Previous research has shown memory complaints are higher in older adults with depression or anxiety versus those without these diagnoses. This suggests that mood symptoms, or a diagnosis of a mood disorder, may represent significant predictors of cognitive impairment. If left untreated, symptoms of depression and memory complaints may lead to greater cognitive impairment, i.e. Mild Cognitive Impairment (MCI) and diagnosis of dementia. Therefore, early interventions are urgently needed to prevent decline in memory and cognitive function in individuals with MCI, depression and/or anxiety.

Ideal interventions for the older aged population would be those that are easily accessible and associated with minimal burden on family members, the healthcare system and the individuals themselves. Mindfulness- Based Stress Reduction (MBSR) therapy and Transcranial Direct Current Stimulation (tDCS) are two interventions that may be effective in targeting cognitive deficits in individuals with anxiety, depression and/ or cognitive complaints. MBSR has been shown to decrease symptoms of depression and improve cognition and tDCS has been shown to improve cognition in the older aged population. The effectiveness of these two interventions combined to elicit changes in cognition has yet to be demonstrated. Therefore, the overall aim of the current research is to evaluate the efficacy of a combination of MBSR and tDCS to improve cognitive function in individuals with anxiety, depression and/or cognitive complaints.

This will be a randomized pilot study. Sixteen individuals (separated into 2 groups of 8) will be randomized to receive a combination of MBSR + active tDCS or MBSR + sham tDCS over 8 weeks. Participants will visit the Healthy Mind Lab once per week for in-class group sessions and will complete the intervention daily at home for the duration of the study. Participants will be aged 60 and older with cognitive complaints, with or without symptoms of anxiety and/or depression. Participants will be trained to self-administer tDCS and given guidelines for the completion of daily MBSR activities at home. It is hypothesized that the combination of active tDCS+MBSR will enhance cognition compared to the combination of sham tDCS + MBSR.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling men and women aged 60 or above.
2. Current cognitive complaints per participant self-report, but with intact cognitive function as defined by a score of 0-9 on the Short Blessed Test (SBT) and a Montreal Cognitive Assessment (MoCA) score ≥25 per PI discretion.
3. PROMIS depression scale score of greater or equal to 16 and/or PROMIS anxiety score greater or equal to 14.
4. Ability to read and speak English fluently enough to complete all research assessments.
5. Corrected visual ability to read newspaper headlines.
6. Hearing capacity to respond to a raised conversational voice.
7. Willingness and ability to provide informed consent.

Exclusion Criteria:

1. The Mini-International Neuropsychiatric Interview (MINI) criteria for current or life-time bipolar disorder, schizophrenia, schizoaffective disorder.
2. Untreated current post-traumatic stress disorder.
3. A MoCA score <25 or SBT score >9, per PI discretion.
4. Use of cognitive enhancers (namely, cholinesterase inhibitors such as donepezil; or memantine) within the past 6 weeks.
5. MINI criteria for any substance abuse within 6 months that would affect their participation, per PI discretion.
6. Unstable medical illness (e.g. uncontrolled diabetes mellitus or hypertension).
7. Concurrent cognitive training, such as brain-training software, participation in psychotherapy or regular engagement in mindfulness practice and/or yoga.
8. Taking anticonvulsant or antipsychotics that cannot be safely tapered and discontinued.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Washington University in Saint Louis, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brooks H, Oughli HA, Kamel L, Subramanian S, Morgan G, Blumberger DM, Kloeckner J, Kumar S, Mulsant BH, Lenze EJ, Rajji TK. Enhancing Cognition in Older Persons with Depression or Anxiety with a Combination of Mindfulness-Based Stress Reduction (MBSR) and Transcranial Direct Current Stimulation (tDCS): Results of a Pilot Randomized Clinical Trial. Mindfulness (N Y). 2021;12(12):3047-3059. doi: 10.1007/s12671-021-01764-9. Epub 2021 Oct 5. PMID 34630733

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham tDCS and MBSR | Active tDCS and MBSR
Started | 14 | 12
Completed | 13 | 10
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham tDCS and MBSR | Active tDCS and MBSR | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (5.0) | 68.3 (5.9) | 68.7 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Cognitive and Memory Function
Description: NIH Toolbox Fluid Cognition Composite Score: provides a global assessment of general fluid cognition functioning. Higher scores indicate higher levels of cognitive functioning. A score at or near 100 indicates ability that is average compared with others nationally. Scores around 115 suggest above-average cognitive ability, while scores around 130 suggest superior ability ( in the top 2 percent nationally). Conversely, a score around 85 suggests below-average cognitive ability and a score in the range of 70 or below suggests significant impairment, which may also be indicative of difficulties in general functioning.
  Fluid abilities are used to solve problems, think and act quickly, and encode new episodic memories. They are presumed to be especially influenced by biological processes and are less dependent on past exposure (learning experiences).
  There is only one primary outcome. No secondary outcomes were reported.
Time Frame: 8 weeks
Population: Twenty-six participants enrolled in the study: 14 were randomized to sham tDCS and 12 to active tDCS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham tDCS and MBSR | Active tDCS and MBSR
Number analyzed (Participants) | 14 | 12
score on a scale | 56.5 (6.7) | 49.8 (7.2)

ADVERSE EVENTS:
Time Frame: Eight weeks
Groups:
- Sham tDCS and MBSR: Includes a combination of 8 weeks of in-class group MBSR + sham tDCS and daily at home MBSR + sham tDCS.
  Sham Transcranial Direct Current Stimulation (tDCS): Transcranial Direct Current Stimulation (tDCS) is a form of neurostimulation (also known as neuromodulation) where very low levels of direct electrical current are delivered to specifically targeted areas of the brain, in order to increase neuroplasticity. The direct current in active tDCS will be of 2 milliampere (mA) (current density = 0.57 A/m2), however, the device is pre-programmed to turn off after 1 minute of active stimulation (and then turn back on briefly at the end of the 30 minutes).
  Most of the adverse events in this study were mild and transient. They included tingling, itching, pain and redness on the scalp, and headaches. Three participants reported worsening of their depressive symptoms; however, this did not lead them to discontinue the study. There were no safety issues associated with tDCS. Adherence with tDCS administration and in-class attendance were comparable in the sham and active groups, suggesting that active tDCS did not cause adverse effects or discomfort associated with non-adherence.
- Active tDCS and MBSR: Includes a combination of 8 weeks of in-class group MBSR + active tDCS and daily at home MBSR + active tDCS.
  Active Transcranial Direct Current Stimulation (tDCS): Transcranial Direct Current Stimulation (tDCS) is a form of neurostimulation (also known as neuromodulation) where very low levels of direct electrical current are delivered to specifically targeted areas of the brain, in order to increase neuroplasticity. The direct current in active tDCS will be of 2 mA (current density = 0.57 A/m2) and will be applied for approximately 30 minutes per day during meditative practices of the MBSR protocol.
  Most of the adverse events in this study were mild and transient. They included tingling, itching, pain and redness on the scalp, and headaches. Three participants reported worsening of their depressive symptoms; however, this did not lead them to discontinue the study. There were no safety issues associated with tDCS. Adherence with tDCS administration and in-class attendance were comparable in the sham and active groups, suggesting that active tDCS did not cause adverse effects or discomfort associated with non-adherence.
Arm/Group | Sham tDCS and MBSR | Active tDCS and MBSR
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 7/14 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham tDCS and MBSR (N=14) | Active tDCS and MBSR (N=12)
Burning and tingling of scalp (Nervous system disorders) | 7 | 6 — Burning and tingling of scalp, itching, headaches associated with electrode placement

LIMITATIONS AND CAVEATS:
Some of the strengths of this feasibility study were a broad range of outcome measures assessing mindfulness, but also cognition, anxiety, depression, and social function; and the length and duration of the tDCS stimulation (10 weeks) that was longer than in most previous studies. The main limitation was the small sample size, which increases the likelihood of both false negative and false positive findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT03653351/Prot_SAP_001.pdf